CLINICAL TRIAL: NCT03982784
Title: Transmuscular Quadratus Lumborum Block for Postoperative Pain After Laparoscopic Partial Nephrectomy: A Randomized Controlled Trial
Brief Title: TQLB for Postoperative Pain After Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: cxl2
Record Dates: First submitted 2019-06-04; First posted 2019-06-12 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Laparoscopic Renal Surgery; Pain Management; Nerve Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-injection TQLB(transmuscular quadratus lumborum block) (Experimental): Single-injection of TQLB is given preoperatively + postoperative IPCA(intravenous patient controlled analgesia)
  Interventions: Procedure: single-injection TQLB(transmuscular quadratus lumborum block); Drug: Morphine given as IPCA(intravenous patient controlled analgesia)
- Control (Active Comparator): postoperative IPCA is given alone
  Interventions: Drug: Morphine given as IPCA(intravenous patient controlled analgesia)

INTERVENTIONS:
Procedure: single-injection TQLB(transmuscular quadratus lumborum block) — Inject 0.6ml/kg local anesthetics in between quadratus lumborum and psoas major under ultrasound guidance
  Arms: single-injection TQLB(transmuscular quadratus lumborum block)
Drug: Morphine given as IPCA(intravenous patient controlled analgesia) — PCIA was initiated using a pump set to deliver boluses of 1.5-2 mg of morphine with a 5-minute lockout interval and no background infusion. The maximal permitted dosage of morphine was set at 8 mg/h.

SUMMARY:
This prospective, randomized study,control study aims to compare the analgesic effect,opioids consumption,quality of recovery,length of hospital stay，et al. between single-injection QLB(quadratus lumborum block)+ intravenous patient-controlled analgesia (IPCA) and intravenous patient-controlled analgesia (IPCA) alone in patients undergoing laparoscopic partial nephrectomy.

ELIGIBILITY:
inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo laparoscopic partial nephrectomy
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption 8 hours after surgery | at the 8 hours after surgery

SECONDARY OUTCOMES:
cumulative morphine consumption at other time points after surgery | at 0, 2, 4, 12, 24 and 48 hours after surgery
The pain scores(at rest or on activity) determined by the numeric rating scale (NRS, 0-10) | at 0, 2, 4, 8,12, 24, 48 and 72 hours after surgery
  NRS is an internationally recognized pain scale with 11 points ranging from 0 to 10 points, with 0 defined as no pain and 10 defined as the worst pain imaginable.
episodes of nausea and vomiting | within 24 hours after the surgery
ambulation time | within the 5 days after surgery
  time from the end of the surgery to the first time to out-of-bed activity
time of recovery of bowl movement | within the 5 days after surgery
  time from the end of the surgery to the first time of bowl movement
patient satisfaction with anesthesia | at 48 hours after surgery
  Patient satisfaction with anesthesia was assessed using a 5-point scale (5: very satisfied; 4: satisfied; 3: neither satisfied nor dissatisfied; 2: dissatisfied; 1: very dissatisfied)
quality of recovery evaluated by the self-assessment 15-item quality of recovery (QoR) scale | at 72 hours and 120 hours after the sugery
  QoR is a 15-item questionnaire which will score on a scale of 0-10 pertaining to patient's comfort, support system, pain, well-being, and ability to carry out daily activities, where 0 indicates none of the time and 10 indicates all of the time
postoperative length of hospital stay | within 2 weeks after the surgery
  time to patient's discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Cui Xulei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided